CLINICAL TRIAL: NCT06792084
Title: The Effect of Motivational Interviewing on Ethical Decision Making and Moral Distress Levels in Intensive Care Nurses: Randomized Controlled Study
Brief Title: The Effect of Motivational Interviewing on Ethical Decision Making and Moral Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nevsehir Haci Bektas Veli University (Other)
Responsible Party: Principal Investigator, Semra seyhan Şahin, RESEARCH ASSISTANT DR, Nevsehir Haci Bektas Veli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NEVU-NRS-SS-01
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Ethics; Moral Distress
Keywords: ethics; moral distress; intensive care nurses
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: It is a pretest-posttest, randomized controlled experimental study with a control group.
Masking Description: There will be no blinding.Randomization will be done to avoid bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participant Information Form, Nursing Ethical Dilemma Test and Moral Distress Scale will be applied to the intervention group to be included in the study before the intervention. Then, the motivational interview program will be implemented in 5 sessions in total, one session per week. At the end of the intervention program, nurses will be asked to fill out the Nursing Ethical Dilemma Test and the Moral Distress Scale.
  Interventions: Behavioral: motivational interviewing
- Control group (No Intervention): No intervention will be applied to the control group to be included in the study. Participants will be asked to fill out the Participant Information Form, Ethical Dilemma Test in Nursing, and Moral Distress Scale forms before and after starting the intervention simultaneously with the intervention group. will be implemented. Then, the motivational interview program will be implemented in 5 sessions in total, one session per week. At the end of the intervention program, nurses will be asked to fill out the Nursing Ethical Dilemma Test and the Moral Distress Scale.

INTERVENTIONS:
Behavioral: motivational interviewing — Motivational interviewing is a directive and client-centered approach used to elicit behavioral change by helping the client explore and resolve ambivalence. Motivational interviewing is a specific method of helping individuals understand their problems and take action for change. In this study, the motivational interview program created in line with the literature (Li et al, 2023; Miller and Rollnick, 2013; Çelik Örücü, 2020) consists of 5 sessions in total, one session per week. There are specific goals and objectives for each session.
  Arms: intervention group

SUMMARY:
The purpose of this study is a pre-test-post-test, randomized controlled experimental study with a control group, planned to examine the effect of motivational interviewing on ethical decision-making and moral distress levels in intensive care nurses.

DETAILED DESCRIPTION:
The research was designed individually. The research will be conducted between 30 JANUARY 2025 and 27 FEBRUARY 2025, with Certificates working in the intensive care units of the Cumhuriyet University Faculty of Medicine in Sivas-Central province of Turkey and meeting the included criteria. The study will be carried out face to face after obtaining the necessary institutional permissions. At each stage of the research, the quantities will be taken into consideration, taking into account the inclusion criteria. They will be asked to fill out informed consent forms asking to explain the subject, purpose and method of receiving the study. Participants will be divided into intervention and control groups by simple randomization method. Participant Information Form, Ethical Dilemma Test in Nursing and Moral Distress Scale will be applied to both groups before the intervention. Data collection tools will be applied to the control group simultaneously with the intervention group. The picture of the implementation of the study will be recorded by the hospital management where appropriate and will be carried out in a private area. At the end of the intervention program, the Nursing Ethical Dilemma Test and Moral Distress Scale will be administered to both groups.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working in Intensive Care Clinics who volunteer to participate in the study will be included.

Exclusion Criteria:

* Being diagnosed with any mental illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Ethical decision making | 5 month
  To reveal the moral problems frequently encountered in patient care; Drawing on her experiences with ethical problems in nursing practice, she developed six dilemmas specific to nursing practice. Principled Thinking demonstrates the importance given to considering moral principles when making moral decisions in nursing. Practical thinking, on the other hand, measures the importance that nurses give to environmental factors such as the number of patients, the number of available resources, institutional policies, the extent to which nurses perceive the support of the management, and physician control, in making decisions regarding ethical issues. The ID and PD scores obtained from each dilemma are added separately to determine the participant's total ID and PD scores. The lowest ID score that can be reached in the test is 18 and the highest ID score is 66. The lowest PD score that can be achieved is 6 and the highest PD score is 36.

SECONDARY OUTCOMES:
Moral Distress | 5 month
  Description: It was developed to evaluate the frequency and intensity of moral distress experienced by nurses working in intensive careThe scale consists of 21 items and consists of 2 dimensions: frequency (0-4) and intensity (0-4). The total score to be obtained from the scale is between 0-336, and an increase in the score indicates an increase in the level of moral distress.

CONTACTS AND LOCATIONS:
Overall Officials: SEMRA SEYHAN ŞAHİN, Dr., Study Director — Nevsehir Haci Bektas Veli University
Locations (1):
- Cumhuriyet University Medical Faculty Hospital, Sivas, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No